CLINICAL TRIAL: NCT06957262
Title: Effects of Surgical Correction of Nasal Obstruction on Oxygen Uptake and Ventilation Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Melekoğlu (Other)
Collaborators: Akdeniz University, Scientific Research Projects Coordination Unit (Unknown)
Responsible Party: Sponsor-Investigator, Tuba Melekoğlu, Assoc. Prof., Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYL-2016-1350
Record Dates: First submitted 2025-04-21; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Nasal Obstruction; Septoplasty Surgeries; Athletic Performance
Keywords: nasal surgery; aerobic performance; exercise economy; respiratory work
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups: an experimental group consisting of athletes with nasal obstruction undergoing septoplasty, and a control group of matched athletes without nasal obstruction who did not receive any intervention. Both groups underwent the same aerobic performance evaluations at baseline and at follow-up (2-3 months).
Masking Description: This study was conducted without masking. Participants and investigators were aware of group assignments due to the nature of the intervention (surgical septoplasty). Outcome assessments (aerobic performance tests and symptom questionnaires) were conducted using objective measures and standardized procedures to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Athletes Undergoing Septoplasty (EG) (Experimental): This arm included male athletes diagnosed with nasal obstruction who underwent surgical correction via septoplasty. Participants were evaluated before and approximately 2-3 months after surgery. Assessments included acoustic rhinometry to measure nasal cavity cross-sectional areas and volumes, the Epworth Sleepiness Scale (ESS), and the Nasal Obstruction Symptom Evaluation (NOSE) scale. Aerobic performance parameters such as running economy, oxygen consumption, and ventilation volume were measured using an incremental treadmill test and respiratory gas analysis.
  Interventions: Procedure: Surgical correction of nasal obstruction
- Control Group (No Intervention): Male athletes without nasal obstruction, matched by age and training level with the experimental group. They did not receive any intervention but underwent the same aerobic performance testing protocol at the same time points for comparison.

INTERVENTIONS:
Procedure: Surgical correction of nasal obstruction — Surgical intervention to correct anatomical nasal obstruction, specifically septal deviation, performed under general anesthesia. The procedure involved the repositioning and reshaping of the deviated nasal septum to improve nasal airflow. The surgery was conducted by an otolaryngologist with experience in nasal airway procedures. No additional medications or postoperative interventions beyond standard care (e.g., saline irrigation, analgesics) were administered. Postoperative assessments occurred 2-3 months after surgery, including evaluations of nasal patency, sleep quality, and aerobic performance using treadmill-based gas exchange measurements.
  Arms: Athletes Undergoing Septoplasty (EG)

SUMMARY:
This retrospective study aims to evaluate the effect of surgical correction of nasal obstruction on aerobic performance parameters in male athletes aged 20-32 years. The main questions it aims to answer are:

* Does nasal obstruction surgery impact running economy and ventilation during exercise?
* Does it affect oxygen consumption during submaximal running efforts?

Researchers will retrospectively compare male athletes who underwent nasal obstruction surgery (experimental group) to matched athletes without nasal obstruction (control group) to assess changes in respiratory function and exercise performance.

Participants were assessed by:

* Acoustic rhinometry to measure nasal cavity dimensions.
* The Nasal Obstruction Symptom Evaluation (NOSE) scale and Epworth Sleepiness Scale (ESS) to evaluate nasal obstruction symptoms and daytime sleepiness.
* Incremental treadmill exercise tests to collect data on gas exchange, oxygen consumption, ventilation, and running economy before and after the surgical intervention (or across a similar time period for the control group).

ELIGIBILITY:
Inclusion Criteria:

For Experimental Group (EG):

* Diagnosed with nasal obstruction due to septal deviation and/or inferior turbinate hypertrophy
* Experiencing nasal breathing difficulties and sleep disturbance
* Deemed eligible for septoplasty and/or inferior turbinoplasty following physical and endoscopic examination
* Voluntarily agreed to participate in the study
* For Control Group (CG):
* No reported nasal obstruction or breathing complications
* Matched with EG participants by age, sport discipline, training level, and VO₂max (with a maximum variation of ±5%)
* Willing to follow a similar training program to their matched EG counterparts between pre- and post-testing periods

Exclusion Criteria:

* History of nasal surgery
* Presence of cardiopulmonary diseases
* Musculoskeletal disorders affecting physical performance or exercise testing
* Inability or unwillingness to follow the pre- and post-test training schedule
* Any surgical complication that would interfere with post-operative participation in physical testing (note: none occurred in this study)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Running Economy (ml/kg/min) | Baseline and 2-3 months post-surgery
  Running economy was assessed via an incremental treadmill test by measuring steady-state oxygen consumption (VO₂) at submaximal running speeds (e.g., 8, 10, 12 km/h). Improvement in running economy is defined by a decrease in VO₂ at the same speed, indicating greater efficiency.

SECONDARY OUTCOMES:
Change in Oxygen Consumption (VO₂ max and submax VO₂) | Baseline and 2-3 months post-surgery
  Peak and submaximal oxygen consumption were evaluated using gas exchange analysis during a graded treadmill test. Reduced submaximal VO₂ values are indicative of improved aerobic performance.
Change in Ventilation | Baseline and 2-3 months post-surgery
  Ventilatory volume was measured during each stage of the treadmill test. Increases in ventilation at submaximal intensities suggest improved airway function and respiratory efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Melekoğlu, Phd, Principal Investigator — Akdeniz University Faculty of Sport Sciences

IPD SHARING:
Plan to Share IPD: Undecided